CLINICAL TRIAL: NCT03844438
Title: A Non-randomized, Open, Dose Escalation Phase 1 Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LPM3480226 Tablets in Patients With Advanced Solid Tumors
Brief Title: A Study Evaluating the Safety, Tolerability of LPM3480226 Tablets in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Luye Pharma Group Ltd. (Industry)
Collaborators: Nanjing Bangnuo Biotechnology Co. Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY01013-CHN -101
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LPM3480226 (Experimental): LPM3480226 tablet will be orally administered，bid，28 days are considered as 1 cycle. The starting dose was 50 mg and the subsequent dose was increased according to the protocol of 100 mg,200 mg,400 mg,600mg.
  Interventions: Drug: LPM3480226

INTERVENTIONS:
Drug: LPM3480226 — The starting dose was 50 mg and the subsequent dose was increased according to the protocol of 100 mg, 200 mg, 400 mg, 600mg.

SUMMARY:
This study is a non-randomized, open, multiple administration and dose escalation phase 1 clinical trial evaluating the safety, tolerability, and pharmacokinetic/pharmacodynamics Characteristics of multiple oral administration of LPM3480226 in patients with advanced solid tumors., determine its dose-limiting toxicity and maximum tolerated dose, and initially observe its clinical effectiveness, and explore the metabolites in plasma after administration.

DETAILED DESCRIPTION:
The primary objective of this study was to assess the safety and tolerability of LPM3480226 tablets after oral administration to patients with advanced solid tumors, and to determine the dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) of LPM3480226.

A non-randomized, open, multiple dose escalation design was used with a total of five dose groups. The starting dose was 50 mg and the subsequent dose was increased according to the protocol of 100 mg , 200 mg , 400 mg , 600mg. Starting from the low-dose group, each subject received only one dose of the drug, and the next dose group study could only be performed if the previous dose group was completed and safe tolerance was confirmed.

Subjects were given the corresponding doses in the order，bid，28 days as a cycle, to evaluate the safety and tolerability of multiple doses. After confirming the safety and tolerance of the dose group in the first administration cycle, the administration was continued for another cycle according to the dose, and the subjects were evaluated for the efficacy after the two-cycle administration, and the subjects who did not have disease progression and is well tolerated and the investigator believes that continued treatment can benefit, the patient may continue to receive the dose of the drug on a voluntary basis, with a maximum dose of no more than one year.

ELIGIBILITY:
Inclusion Criteria:

* The subject has voluntarily signed the written informed consent form (ICF)
* Male or female patients aged 18 to 75 years (18 years and 75 years are inclusive)
* Advanced solid tumors confirmed by histology or cytology (the following tumors may be preferred: melanoma, bladder cancer, kidney cancer, head and neck cancer, lung cancer, etc.);
* Standard treatment is ineffective, subjects refuse to accept or cannot tolerate standard treatment, or there is no standard effective treatment;
* The patient should have at least one measurable lesion as the target lesion (according to RECIST 1.1 criteria)
* The Eastern Cooperative Oncology Group (ECOG) performance status score is < 2 point.
* The predictable survival duration is ≥ 3 months
* Laboratory results during screening: absolute neutrophil count ≥ 1.5× 109/L; platelet count≥ 90× 109/L; hemoglobin≥ 90 g/L; Total bilirubin ≤1.5×upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2.5×ULN for the subjects without liver metastasis and ALT and AST< 5×ULN for the subjects with liver metastasis.; creatinine clearance ≥ 50 mL/min （Cockcroft-Gault formula)
* QTc interval male ≤ 450 ms female≤ 470 ms；
* The female subjects and male subjects of childbearing age and the partners of the male subjects agree to take reliable contraceptive measures during the study period and within 6 months after infusion of the study drugs

Exclusion Criteria:

* There are any active autoimmune diseases or a history of autoimmune diseases [including but not limited to: rheumatoid arthritis, ankylosing spondylitis, autoimmune hemolytic anemia, interstitial pneumonia, uveitis, inflammation Intestinal disease, autoimmune hepatitis, autoimmune hypophysitis, glomerulonephritis, hyperthyroidism or decreased thyroid function (subclinical patients can be included), allergic asthma (where asthma in childhood has been completely relieved, and no intervention needed in adults can be included. Patients with asthma who need bronchodilators for medical intervention cannot be included.), and patients with vitiligo and type 1 diabetes can be included];
* Brain metastases, spinal cord compression, or cancerous meningitis, or brain CT or MRI scans confirmed brain metastases during screening period;
* have gastrointestinal diseases that may affect the absorption of the drug, or have undergone gastrointestinal surgery, which may affect the drug absorption by the investigator;
* Previously received radiotherapy, chemotherapy, surgery, or small molecule targeted therapy, less than 4 weeks prior to the first dose after treatment (if you had previously received nitrosourea or mitomycin chemotherapy, the time between the end of chemotherapy and the first dose Less than 6 weeks);
* Continue to use immunosuppressants (including but not limited to: tacrolimus, cyclosporine, etc.), systemic or topical hormonal therapy (dose > 10 mg / day prednisone or corresponding equivalent of other hormones)within 2 weeks prior to the first dose;
* Those who have received any vaccine within 28 days prior to the first dose;
* Any drug that affects tryptophan metabolism is used within 28 days prior to the first dose, including but not limited to: serotonin reuptake inhibitors (eg, fluoxetine, paroxetine, fluvoxamine, sertraline, Citalopram, escitalopram, etc.), tryptophan hydroxylase inhibitors (eg, trossostat ethyl ester, p-chlorophenylalanine, etc.);
* Those who have used CYP3A4 strong inducers or strong inhibitors within 2 weeks before the first dose or within 5 half-life periods (for long periods of time) (see Annex V);
* Immunological "checkpoint" inhibitors (including but not limited to: anti-PD-1/PD-L1/PD-L2 monoclonal antibodies, anti-CTLA-4 monoclonal antibodies) were used within 42 days prior to the first dose;
* A monoamine oxidase inhibitor or a drug having a monoamine oxidase inhibitory action (eg, pethidine hydrochloride, linezolid, methylene blue, etc.) is used 3 weeks before the first administration or within 5 half-life periods (for long periods of time);
* Interferon-treated within 6 months prior to the first dose;
* Those who have used IDO/TDO inhibitors in the past;
* Active infections;
* Any of Hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibody (HCV-Ab), acquired immunodeficiency syndrome antibody (Anti-HIV) or treponema pallidum antibody (TP-Ab) is positive;
* Those who received any other study drug or participated in another interventional clinical study 28 days before the first dose (42 days for mAbs);
* Other systemic anti-tumor therapists may be accepted during the study;
* Known to have a history of psychotropic substance abuse, alcohol abuse or drug abuse;
* Pregnant, lactating women or women with fertility test positive for pregnancy test;
* other important organ primary diseases (such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system or metabolic endocrine system disease) or other reasons which are considered by the investigator that the subject is unsuitable to be enrolled.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-12-18 (Actual); Primary Completion 2020-10-28 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of LPM3480226 assessed by adverse events | 1 cycle (28 days)
  Collection of adverse events throughout the study as a measure of safety and tolerability.

SECONDARY OUTCOMES:
AUC | 1 cycle (28 days)
  Area under the concentration-time curve (AUC) Assessment Area under the concentration-time curve (AUC) for the Pharmacokinetics (PK) of
CMax | 1 cycle (28 days)
  Maximum concentration (Cmax) Assessment Maximum concentration (Cmax) for the Pharmacokinetics (PK) of

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Zoubi RM, Elaarag M, Al-Qudimat AR, Al-Hurani EA, Fares ZE, Farhan A, Al-Zoubi SR, Khan A, Agouni A, Shkoor M, Bawadi H, Zakaria ZZ, Al Zoubi M, Alrumaihi K. IDO and TDO inhibitors in cancer immunotherapy: mechanisms, clinical development, and future directions. Front Pharmacol. 2025 Sep 16;16:1632446. doi: 10.3389/fphar.2025.1632446. eCollection 2025. PMID 41035912